CLINICAL TRIAL: NCT00923624
Title: Patient Portal to Support Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01MH081750 (NIH); 5R01MH081750 (NIH)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Antiretroviral Medication Adherence
Keywords: electronic medical record; antiretroviral medication adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- staff emails (Active Comparator): Attention control that includes staff sending emails with information about using health information technology system.
  Interventions: Other: attention control
- study nurse messages (Experimental): A series of 6 proactive secure messages and 3 proactive booster messages (for a total of 9 secure and personalized messages) sent by the study nurse via the EMR patient web portal.
  Interventions: Behavioral: adherence intervention

INTERVENTIONS:
Other: attention control — 9 informational email messages sent by study staff about the features of the shared electronic medical record system and how to use them.
  Arms: staff emails
Behavioral: adherence intervention — 9 messages tailored by the study nurse and guided by the IMB model
  Arms: study nurse messages

SUMMARY:
The purpose of this study is to conduct a randomized control trial of a behavioral intervention delivered by nurses via an electronic medical record (EMR) patient web portal to determine if this is an efficacious method for supporting medication adherence.

DETAILED DESCRIPTION:
300 adult HIV+ patients will be randomized to one of two arms. 150 will be assigned to receive secure messages focused on antiretroviral adherence from a nurse through the health plan EMR patient website. 150 will be assigned to an attention control comparison arm, and will receive electronic messages from a study staff member that provide information about the various features of the health plan patient website. Patients will be invited by mail to be telephone screened for enrollment in the study. Patients will be provided the opportunity to opt out of being contacted by the study. Eligible and interested patients will be mailed an access code and separately emailed a link to a secure study website where they will complete a web consent form and a baseline web survey before being randomized to an intervention arm. This trial will allow us to evaluate the effectiveness of using health information technology as an intervention delivery vehicle to improve patient disease management behaviors such as treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in GHC or KP health plans for at least 6 months
* expect to stay enrolled for 1 year in health plan
* HIV+
* currently prescribed antiretroviral medication
* regular access to a computer with internet capabilities and working email address and meet one of the following:
* gap in antiretroviral prescription refills based on 6 month refill records
* referral to study by provider team for adherence problems

Exclusion Criteria:

* dementia or psychosis diagnosis documented in medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Lapses in medication adherence over the last 7 and 30 days (self report) and over previous 12 months (pharmacy records). | 12 months

SECONDARY OUTCOMES:
Web service utilization. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl L. Catz, PhD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Oakland, California
  - Group Health Research Institute, Seattle, Washington